CLINICAL TRIAL: NCT04249583
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of QM1114-DP for the Treatment of Moderate to Severe Glabellar Lines
Brief Title: Treatment of Moderate to Severe Glabellar Lines
Acronym: READY-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 43QM1602
Record Dates: First submitted 2019-12-30; First posted 2020-01-31 (Actual); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2022-09

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): QM1114-DP, a Botulinum Toxin Type A (BoNT-A) ; Mode of administration: intramuscular injection
  Interventions: Biological: botulinum toxin
- Placebo (Placebo Comparator): A buffered solution; Mode of administration: intramuscular injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: botulinum toxin — neuromodulator to be injected in the GL region
  Other Names: QM1114-DP
  Arms: Treatment
Biological: Placebo — Placebo to be injected in the GL area
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate the efficacy and safety of a single dose of QM1114-DP compared to placebo for the treatment of moderate to severe GL.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age or older.
2. Moderate to severe GL at maximum frown as assessed by the Investigator.
3. Moderate to severe GL at maximum frown as assessed by the subject.

Exclusion Criteria:

1. Previous use of any Botulinum toxin in facial areas within 9 months prior to study treatment.
2. Female who is pregnant, breast feeding, or intends to conceive a child during the study.
3. Known allergy or hypersensitivity to any component of the investigational product (QM1114-DP) or any botulinum toxin serotype.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2021-01-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (13):
  - \Ablon Skin Institute and Research Center, Manhattan Beach, California
  - Moradi MD, Vista, California
  - Etre Cosmetic Dermatology and Laser Center, New Orleans, Louisiana
  - Maryland Dermatology, Laser Skin & Vein, Hunt Valley, Maryland
  - Skin Specialist, PC, Omaha, Nebraska
  - Robert Schwarcz, MD, PC, New York, New York
  - Sachin M Shridharani, MD, New York, New York
  - Wilmington Dermatology Center, PLLC, Wilmington, North Carolina
  - The Practice of Brian S Biesman, MD, Nashville, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Dallas Center for Dermatology & Aesthetics, Dallas, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - Integrated Aesthetics, Inc, Spring, Texas
- Sweat Clinics of Canada, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 225 | 75
Completed | 210 | 66
Not Completed | 15 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 223 | 74 | 297
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (12.41) | 47.6 (11.19) | 47.6 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 203 | 65 | 268
  Male | 20 | 9 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 4
  Asian | 8 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 7 | 24
  White | 185 | 61 | 246
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With a ≥ 2-grade Improvement From Baseline on the Glabellar Lines Investigator and Subject Assessments at Maximum Frown at One Month.
Description: The investigator and subject evaluate the subject's GL severity using a 4-grade scale (0 = none and 3 = severe)
Time Frame: One Month
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 199 | 67
Participants | 165 | 0
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.05, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percentage of Subjects With a 0 or 1 on the Glabellar Lines Investigator Scale at Maximum Frown
Time Frame: One Month
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 194 | 64
Participants | 187 | 3

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/222 | 0/75
Serious Adverse Events (participants affected / at risk) | 5/222 | 1/75
Other Adverse Events (participants affected / at risk) | 8/222 | 2/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=222) | Placebo (N=75)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=222) | Placebo (N=75)
COVID-19 (Infections and infestations) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/83/NCT04249583/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT04249583/SAP_001.pdf